CLINICAL TRIAL: NCT02632916
Title: A Single-Blinded, Randomized, Controlled, Phase 2 Pilot Study to Evaluate the Safety and Efficacy of Denosumab Compared to Zoledronic Acid for the Treatment of Osteoporosis in Children
Brief Title: Denosumab for the Treatment of Osteoporosis in Children: A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Dr. Leanne Ward, MD, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DZA9DEC2015
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid; Denosumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Zoledronic Acid (Active Comparator): Intravenous zoledronic acid 0.025mg/kg
  Interventions: Drug: Zoledronic Acid
- Denosumab (Experimental): Subcutaneous denosumab 1.0mg/kg
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Zoledronic Acid — Intravenous zoledronic acid 0.025mg/kg at baseline, 6 months, 12 months and 18 months
  Arms: Zoledronic Acid
Drug: Denosumab — Subcutaneous denosumab 1.0mg/kg at baseline, 6 months, 12 months and 18 months
  Arms: Denosumab

SUMMARY:
The aim of this study is to acquire preliminary, pilot data over a 2-year period on the safety and efficacy of subcutaneous denosumab versus the current CHEO standard-of-care (intravenous zoledronic acid) for the treatment of osteoporosis in children. Both denosumab (1.0mg/kg) and zoledronic acid (0.025mg/kg) will be given as four doses separated by a six month interval (i.e. at baseline, 6 months, 12 months and 18 months), with follow-up to 2 years.

DETAILED DESCRIPTION:
Bone fractures without significant trauma (also known as osteoporosis) are a frequent complication of chronic childhood diseases (for example, Duchenne muscular dystrophy and inflammatory disorders) and genetic disorders (such as osteogenesis imperfecta). To date, the only effective therapy for the treatment of osteoporosis in children is a class of medications known as bisphosphonates (which include pamidronate and zoledronic acid). Unfortunately, these medications have the disadvantage of frequent side effects with the first dose (including fever, nausea, vomiting and bone pain), as well as intravenous administration (delivery through a vein, similar to a bloodtest). Recently, a new medication has been proven effective in the treatment of adults with osteoporosis - this medication is called denosumab, and it has a distinct advantage over intravenous bisphosphonates since it is administered sub-cutaneously (through a small needle injected into the skin), plus an excellent safety profile. To date, denosumab has been used with success in a few children with rare forms of osteoporosis and other bone disorders. The purpose of this study is to further test the safety and benefits of denosumab in children with fractures due to osteoporosis, by comparing this new agent to the current standard treatment at CHEO, zoledronic acid. This will be a one year, pilot study in 20 children with a variety of forms of osteoporosis. Children enrolled in the study will be randomly assigned to receive zoledronic acid or denosumab every 6 months (for two doses), with tests carried out every few months over the course of the year to study the effects of these therapies on fractures, bone density and various safety parameters as measured by bloodtests. Overall, the results of this study will provide us with important information on the potential for denosumab to provide children with a safe, effective and convenient new osteoporosis treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's legally acceptable representative has provided informed consent.
2. Children aged 4 to 16 years at the time of enrolment.
3. Children with a history of clinically significant bone fragility in the preceding 24 months, requiring the child to have ONE or more of the following clinical profiles:

   1. At least one low-trauma vertebral or long bone fracture in a child with an underlying disease known to be associated with osteoporotic fractures (e.g. glucocorticoid-treated diseases, Crohn's disease, rheumatic disorders, Duchenne muscular dystrophy, other muscular dystrophies, spinal muscular atrophy, cerebral palsy); OR
   2. At least one low-trauma vertebral or long bone fracture in the last 24 months, in a child with a known genetic osteoporotic condition such as osteogenesis imperfecta (confirmed on molecular genetic testing); OR
   3. At least one low-trauma vertebral or long bone fracture in the last 24 months, in an otherwise healthy child with a diagnosis of osteoporosis confirmed on trans-iliac bone biopsy. Trans-iliac bone biopsy is a requirement in this sub-group as per the usual standard of care, as this is the only test that will definitively confirm osteoporosis in an otherwise healthy child who does not have a genetic bone fragility condition.

Exclusion Criteria:

1. Any child for whom the treating physician feels participation is not advised.
2. Prior treatment with an osteoporosis agent (e.g. bisphosphonate).
3. Renal insufficiency defined as an eGFR less than 60ml/min/1.73m2.
4. Active or prior diagnosis of malignancy or undergoing investigations for a suspected childhood cancer.
5. Currently breastfeeding or plans to breastfeed during the study.
6. Pregnancy (verified by pre-treatment pregnancy test in all menstruating or sexually active females).
7. Untreated vitamin D deficiency, defined as a serum 25OHD level <50nmol/L.
8. Untreated hypocalcemia, defined as a serum ionized calcium level <1.1mmol/L.
9. Active or historic eczema/cellulitis.
10. Children planning dental procedures and/or dental surgery during the course of the study.
11. Children with a documented history of atrial fibrillation.
12. Children with asthma who are acetylsalicylic acid (ASA) sensitive.
13. Children that have had parathyroid or thyroid surgery.
14. Children who are allergic to rubber or latex.
15. Males with a pregnant partner.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
The changes in serum ionized calcium levels at 48 hours following the administration of denosumab versus zoledronic acid. | 48 hours after each drug administration (48 hours post baseline and 48 hours post 6, 12 and 18 month visits)
  To observe the changes in serum ionized calcium levels at 48 hours following the administration of denosumab versus zoledronic acid. Hypocalcemia at 48 hours has been chosen as the primary outcome since this is a clinically important side effect of both denosumab and zoledronic acid, and 48 hours is around the time of the anticipated calcium nadir

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Ward, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
No current plan
Time Frame: No time frame
Access Criteria: Access has not been made available